CLINICAL TRIAL: NCT02022826
Title: Clinical Management With SmartPill Motility Monitoring System and Validation of the SmartPill Five Hour Cutoff in Patients With Symptoms of Gastroparesis
Brief Title: Clinical Management With SPM System and Validation of the SPM 5 Hour Cutoff in Patients With Symptoms of Gastroparesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor internal decision
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-501
Record Dates: First submitted 2013-12-15; First posted 2013-12-30 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-08

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; SmartPill Monitoring System (SPM); Gastric Emptying Scintigraphy (GES)
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SmartPill Monitoring System (Experimental): patients with symptoms of Gastroparesis will undergo the SmartPill monitoring system test
  Interventions: Device: SmartPill Monitoring System

INTERVENTIONS:
Device: SmartPill Monitoring System
  Other Names: SPM

SUMMARY:
This protocol is designed to validate use of the SPM for diagnosis of delayed gastric emptying in patients with symptoms of gastroparesis and assess impact of a SmartPill study on patient management in the gastroparetic populations. Patients with symptoms of gastroparesis will be recruited.

Patients will undergo concurrent gastric scintigraphy and SPM testing to determine the presence or absence of delayed gastric emptying based on predetermined diagnostic cutoffs for each technique.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages of 18-80 years of age with symptoms of gastroparesis for at least 12 weeks.
* Presenting with 2 or more of the following symptoms or signs which, in the opinion of the site investigator, are suggestive of a diagnosis of gastroparesis:

  * 1 Nausea, vomiting, or retching (dry heaves)
  * 2 Postprandial fullness or early satiety
  * 3 Bloating or visible abdominal distention
  * 4 Postprandial discomfort or pain
* Ability to stop proton pump inhibitors for 7 days and histamine2 receptor antagonists, prokinetic agents, narcotic agents, anticholinergic drugs, and cannabinoids 3 days prior to SPM and gastric scintigraphy testing.
* No evidence of metabolic disease (hypothyroidism, uncontrolled diabetes [hemoglobin A1c >10% within the past 6 months], electrolyte imbalance).
* An upper endoscopy or upper gastrointestinal barium series within the past 2 years showing no organic disease that is potentially causative of symptoms.
* High probability of compliance and completion of study.

Exclusion Criteria:

* Participation in previous SmartPill clinical trials.
* Previous history of bezoars (the presence of retained liquid, bile, or small amounts of poorly organized food residue is permitted).
* Dysphagia to solid food or pills.
* Prior surgery involving the luminal gastrointestinal tract (cholecystectomy, appendectomy, and hysterectomy are permitted if performed > 3 months prior to SPM test).
* Any abdominal or pelvic surgery within the past 3 months
* Known or history of inflammatory bowel disease.
* History of diverticulitis, diverticular stricture, and other intestinal strictures.
* Chronic daily use of nonsteroidal anti-inflammatory drugs (ibuprofen, naproxen, etc.)
* Tobacco or alcohol use within eight hours prior to capsule ingestion.
* BMI > 40 kg/m2.
* Allergies to eggs, bread, or jam.
* Females of childbearing age who are not practicing birth control and/or are pregnant or lactating. (Urine pregnancy testing will be performed on female subjects of child-bearing potential prior to capsule ingestion and gastric scintigraphy).
* Use of cardiac medical devices such as pacemakers and defibrillators (gastric stimulators, bladder stimulators, spinal stimulators, medication infusion devices, insulin pumps, continuous glucose monitors are permitted).
* Uncontrolled diabetes with a hemoglobin A1c >10%.
* Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Braden Kuo, Dr., Principal Investigator
Locations (11):
- United States (11):
  - Stanford University, Palo Alto, California
  - Florida Digestive Health, Largo, Florida
  - Miami miller school of Medicin, Miami, Florida
  - Georgia Regents University, Augusta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Temple University, Philadelphia, Pennsylvania
  - Clinsearch,LLC, Chattanooga, Tennessee
  - Texas Tech University, El Paso, Texas
  - Fletcher Allen Health Care, Burlington, Vermont

REFERENCES:
- [Derived] Surjanhata BC, Moshiree B, Lee AA, McCallum RW, Sarosiek I, Nguyen LA, Schulman MI, Wo JM, Parkman HP, Kuo B, Hasler WL, Rao SSC. Impact of Constipation Therapies on Severity of Gastroparesis and Constipation Symptoms in Relation to Gastric and Colonic Transit. Neurogastroenterol Motil. 2025 Jun;37(6):e70013. doi: 10.1111/nmo.70013. Epub 2025 Mar 3. PMID 40033166
- [Derived] Hasler WL, Lee AA, Moshiree B, Surjanhata BC, Rao S, Parkman HP, Nguyen LA, Sarosiek I, Wo JM, Schulman MI, McCallum RW, Kuo B. Benefits of Prokinetics, Gastroparesis Diet, or Neuromodulators Alone or in Combination for Symptoms of Gastroparesis. Clin Gastroenterol Hepatol. 2024 Apr;22(4):867-877.e12. doi: 10.1016/j.cgh.2023.10.014. Epub 2023 Oct 30. PMID 37913936
- [Derived] Lee AA, Rao K, Parkman HP, McCallum RW, Sarosiek I, Nguyen LA, Wo JM, Schulman MI, Moshiree B, Rao S, Kuo B, Hasler WL. Baseline Predictors of Longitudinal Changes in Symptom Severity and Quality of Life in Patients With Suspected Gastroparesis. Clin Gastroenterol Hepatol. 2022 Mar;20(3):e407-e428. doi: 10.1016/j.cgh.2020.09.032. Epub 2020 Sep 21. PMID 32971231
- [Derived] Hasler WL, Rao SSC, McCallum RW, Krause RA, Nguyen LA, Schulman MI, Lee AA, Moshiree B, Wo JM, Parkman HP, Sarosiek I, Wilding GE, Kuo B. Influence of Gastric Emptying and Gut Transit Testing on Clinical Management Decisions in Suspected Gastroparesis. Clin Transl Gastroenterol. 2019 Oct;10(10):e00084. doi: 10.14309/ctg.0000000000000084. PMID 31663906
- [Derived] Lee AA, Rao S, Nguyen LA, Moshiree B, Sarosiek I, Schulman MI, Wo JM, Parkman HP, Wilding GE, McCallum RW, Hasler WL, Kuo B. Validation of Diagnostic and Performance Characteristics of the Wireless Motility Capsule in Patients With Suspected Gastroparesis. Clin Gastroenterol Hepatol. 2019 Aug;17(9):1770-1779.e2. doi: 10.1016/j.cgh.2018.11.063. Epub 2018 Dec 14. PMID 30557741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period- January 2014 March 2017; 11 academic and community centers within the US
Pre-assignment Details: medication wash out period: Subjects instructed to discontinue agents that affect intragastric acidity including proton pump inhibitors for 7 days, histamine2 receptor antagonists for 3 days and antacids for 1 day prior to study including the day of SPM ingestion.
Period: Overall Study
Arm/Group | SmartPill Monitoring System
Started | 167
Completed | 139
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | SmartPill Monitoring System
Number analyzed (Participants) | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 154
  >=65 years | 13
Age, Continuous [Mean (Full Range); unit: years] | 45 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 167
suspected gastroparesis [Count of Participants; unit: Participants] | 167

OUTCOME MEASURES:

1. Primary Outcome: Per Patient Device Agreement Between SmartPill Motility Monitoring System Gastric Emptying Time & Gastric Emptying Scintigraphy Test in Patients With Symptoms of Gastroparesis
Description: Per patient device agreement for the diagnosis of delayed gastric emptying between SmartPill Motility Monitoring System (SPM) gastric emptying time (GET >5 hours) and the non-reference standard, gastric Emptying scintigraphy test (>10% retention of a solid meal at 4 hours) in patients with symptoms of gastroparesis
Time Frame: an expected average of two weeks from study procedure
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | SmartPill Monitoring System
Number analyzed (Participants) | 152
percentage of agreement | 76 [69 to 83]
Statistical Analysis 1: Comparison: SmartPill Monitoring System; Test type: Other; p = 0.0052, McNemar; percentage of agreement = 76, 95% CI 2-sided [69 to 83]

2. Secondary Outcome: Agreement Between Gastric Emptying Time of SmartPill Capsule and Gastroduodenal Contractility and Percent of Radiolabeled Meal Retained at 4 Hours on Scintigraphy for Severe Gastroparesis
Description: Agreement between Gastric emptying time of SmartPill capsule (GET>8hrs= severe) and gastroduodenal contractility and percent of radiolabeled meal retained at 4 hours on scintigraphy (>35% = severe)
Time Frame: an expected average of two weeks from study procedure
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | SmartPill Monitoring System
Number analyzed (Participants) | 143
percentage of agreement | 92 [87 to 96]
Statistical Analysis 1: Comparison: SmartPill Monitoring System; Test type: Other; p = 1.00, McNemar; precentage of agreement = 92, 95% CI 2-sided [87 to 96]

ADVERSE EVENTS:
Time Frame: Adverse events collected from beginning of enrollment to last patient last visits: January 2014-March 2017 (2 years and 3 months)
Arm/Group | SmartPill Monitoring System
All-Cause Mortality (participants affected / at risk) | 2/167
Serious Adverse Events (participants affected / at risk) | 10/167
Other Adverse Events (participants affected / at risk) | 18/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartPill Monitoring System (N=167)
Nausea and Vomiting (Gastrointestinal disorders) | 4 (5)
dehydration (General disorders) | 1 (1)
uncontrolled high blood pressure (Blood and lymphatic system disorders) | 1 (1)
exacerbation of pre-existing condition secondary to gastroparesis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
kidney translant (Renal and urinary disorders) | 1 (1)
capsule retention (Gastrointestinal disorders) | 1 (1)
laproscopic-assisted vaginal historectomy and right salpingo-oophorectomy (Reproductive system and breast disorders) | 1 (1)
Right Hip Replacement (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartPill Monitoring System (N=167)
Abdominal Pain (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dumping syndrome (Gastrointestinal disorders) | 1 (1) — Dumping syndrome
kidney translant (Reproductive system and breast disorders) | 3 (4) — pregnancy
Brain Aneurysm (Nervous system disorders) | 1 (1) — Brain Aneurysm
extreme pain and bloating (Gastrointestinal disorders) | 1 (1) — extreme pain and bloating
Right Hip Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) — body aches and arthralgia
Upper Respitory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Upper Respiratory Infection
labioplasty with bilateral simple partial vulvectomy (Reproductive system and breast disorders) | 1 (1) — labioplasty with bilateral simple partial vulvectomy
facial droop, ER visit; diagnosed with Bell's palsy (Nervous system disorders) | 1 (1) — facial droop, ER visit; diagnosed with Bell's palsy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-03-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT02022826/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02022826/SAP_001.pdf